CLINICAL TRIAL: NCT01864785
Title: Posterior Fixation Alone Versus Posterior Fixation Combined With Articular Process Fusion in Thoracolumbar Burst Fractures
Brief Title: Comparison of Posterior Fixation Alone and Combined With Articular Process Fusion in Thoracolumbar Burst Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Zhonghua Ling, resident, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xblzh2013
Record Dates: First submitted 2013-05-19; First posted 2013-05-30 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Thoracolumbar Burst Fracture
Keywords: Operative treatment; internal fixation; posterior spinal fusion
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixation Alone (Other): Use the Posterior approach to achieve the reduction and stabilization by pedicle screw and rod alone
  Interventions: Procedure: Fixation Combined With Fusion
- Fixation Combined With Fusion (Other): Posterior Fixation Combined With Articular Process Fusion in thoracolumbar Fracture.
  Interventions: Procedure: Fixation Alone

INTERVENTIONS:
Procedure: Fixation Combined With Fusion — Articular process fusion with bone graft was carried out after screw fixation
  Arms: Fixation Alone
Procedure: Fixation Alone — Use the Posterior approach to achieve the reduction and stabilization by pedicle screw and rod alone
  Arms: Fixation Combined With Fusion

SUMMARY:
Nearly 90% of all spinal fractures occur in the thoracolumbar region, and burst fractures are composed of 15% of such injuries. But the treatment of thoracolumbar fractures remains controversial. Treatment varies from the conservative management to various types of surgery. Internal fixation with spinal fusion is a surgical treatment method that is generally accepted for patients with thoracolumbar fracture. In this department, the investigators treat thoracolumbar burst fracture with posterior fixation alone and combined with articular process fusion. To evaluate the result of the two kinds of treatment, the investigators design this clinical trial. So, the investigators compared the radiological and clinical outcomes between patients who underwent posterior fixation alone and supplemented with fusion following the onset of thoracolumbar burst fractures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of thoracolumbar burst fracture

Exclusion Criteria:

* smoking during the period of the trial
* conservative treatment could be attempted
* do not meet the requirements of follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Cobb angle | 3 days after surgery.
  Cobb angle is a variable for kyphotic deformity assessment
Cobb angle | 3 months after surgery
  Cobb angle is a variable for kyphotic deformity assessment
Cobb angle | 12 months after surgery
  Cobb angle is a variable for kyphotic deformity assessment
Cobb angle | 18 months after surgery
  Cobb angle is a variable for kyphotic deformity assessment

SECONDARY OUTCOMES:
failure of internal fixation | 3days after surgery
failure of internal fixation | 3 months after surgery
failure of internal fixation | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xu bin, master, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Ghobrial GM, Jallo J. Thoracolumbar spine trauma: review of the evidence. J Neurosurg Sci. 2013 Jun;57(2):115-22. PMID 23676860
- [Result] Hwang JU, Hur JW, Lee JW, Kwon KY, Lee HK. Comparison of posterior fixation alone and supplementation with posterolateral fusion in thoracolumbar burst fractures. J Korean Neurosurg Soc. 2012 Oct;52(4):346-52. doi: 10.3340/jkns.2012.52.4.346. Epub 2012 Oct 22. PMID 23133723
- [Result] Jindal N, Sankhala SS, Bachhal V. The role of fusion in the management of burst fractures of the thoracolumbar spine treated by short segment pedicle screw fixation: a prospective randomised trial. J Bone Joint Surg Br. 2012 Aug;94(8):1101-6. doi: 10.1302/0301-620X.94B8.28311. PMID 22844053
- [Result] Islam MA, Sakeb N, Islam A, Sarker SK, Mondol SK. Evaluation of the results of posterior decompression, posterolateral fusion and stabilization by pedicle screw and rod in traumatic thoracolumbar fractures. Bangladesh Med Res Counc Bull. 2011 Dec;37(3):97-101. doi: 10.3329/bmrcb.v37i3.9121. PMID 22352229
- [Result] Schmid R, Lindtner RA, Lill M, Blauth M, Krappinger D, Kammerlander C. Combined posteroanterior fusion versus transforaminal lumbar interbody fusion (TLIF) in thoracolumbar burst fractures. Injury. 2012 Apr;43(4):475-9. doi: 10.1016/j.injury.2011.12.011. Epub 2012 Jan 9. PMID 22227107
- [Result] Ge CM, Wang YR, Jiang SD, Jiang LS. Thoracolumbar burst fractures with a neurological deficit treated with posterior decompression and interlaminar fusion. Eur Spine J. 2011 Dec;20(12):2195-201. doi: 10.1007/s00586-011-1875-6. Epub 2011 Jun 18. PMID 21688000